CLINICAL TRIAL: NCT01167881
Title: A Phase III Randomised, Double-blind, Active-controlled Parallel Group Efficacy and Safety Study of BI 10773 Compared to Glimepiride Administered Orally During 104 Weeks With a 104 Week Extension Period in Patients With Type 2 Diabetes Mellitus and Insufficient Glycaemic Control Despite Metformin Treatment
Brief Title: Efficacy and Safety of Empagliflozin (BI 10773) With Metformin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.28; 2009-016244-39 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-07-15; First posted 2010-07-22 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; glimepiride

ARMS (2):
- BI 10773 dose plus metformin (Experimental): Patients receive one BI10773 tablet and one placebo Glimepiride capsule once daily
  Interventions: Drug: BI 10773; Drug: Placebo
- Glimepiride 1-4 mg plus metformin (Active Comparator): Patients receive one glimepiride capsule and one placebo tablet Bi 10773 once daily.
  Interventions: Drug: Glimepiride; Drug: Placebo

INTERVENTIONS:
Drug: BI 10773 — Medium dose once daily
  Arms: BI 10773 dose plus metformin
Drug: Glimepiride — 1-4 mg once daily
  Arms: Glimepiride 1-4 mg plus metformin
Drug: Placebo — Placebo matching BI 10773
  Arms: Glimepiride 1-4 mg plus metformin
Drug: Placebo — Placebo matching Glimepiride
  Arms: BI 10773 dose plus metformin

SUMMARY:
This is a pivotal phase III study, mandatory to seek approval by regulatory authorities for BI 10773 as an anti-diabetic agent compared to an active comparator in patients with type 2 diabetes mellitus and insufficient glycaemic control.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis typ 2 diabetes mellitus
* Male and female on diet and exercise regimen, pre-treated with metformin 12 weeks prior to randomisation
* HbA1c equal or greater than 7.0% and less than or equal to 10% at visit 1
* 18 years or more
* BMI equal or less than 45Kg/m2

Exclusion criteria:

* Uncontrolled hyperglycemia defined as glucose more that 13.3 mmol/L after overnight fast during placebo run-in
* Any other antidiabetic drug within 12 weeks prior to randomisation except metformin
* Acute coronary syndrome (non-STEMI, STEMI unstable angina pectoris), stroke or transient ischemic attack within 12 weeks of informed consent
* Indication of liver disease
* Moderate to severe renal impairment
* Bariatric surgery within past 2 years
* Medical history of cancer or treatment for cancer within last 5 years
* Blood dyscrasias or any disorders causing haemolysis or unstable red blood cell
* Contraindications hypersensitivity to concomitant drugs
* Treatment with anti-obesity drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1549 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (182):
- United States (25):
  - 1245.28.10005 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1245.28.10012 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1245.28.10016 Boehringer Ingelheim Investigational Site, Hot Springs, Arkansas
  - 1245.28.10003 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 1245.28.10021 Boehringer Ingelheim Investigational Site, West Hills, California
  - 1245.28.10009 Boehringer Ingelheim Investigational Site, Bradednton, Florida
  - 1245.28.10015 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1245.28.10033 Boehringer Ingelheim Investigational Site, Blue Ridge, Georgia
  - 1245.28.10026 Boehringer Ingelheim Investigational Site, Boise, Idaho
  - 1245.28.10007 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1245.28.10027 Boehringer Ingelheim Investigational Site, Henderson, Nevada
  - 1245.28.10014 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 1245.28.10006 Boehringer Ingelheim Investigational Site, Shelby, North Carolina
  - 1245.28.10011 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1245.28.10019 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1245.28.10004 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1245.28.10008 Boehringer Ingelheim Investigational Site, Perrysburg, Ohio
  - 1245.28.10020 Boehringer Ingelheim Investigational Site, Medford, Oregon
  - 1245.28.10017 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1245.28.10031 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1245.28.10032 Boehringer Ingelheim Investigational Site, Longview, Texas
  - 1245.28.10022 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1245.28.10030 Boehringer Ingelheim Investigational Site, Draper, Utah
  - 1245.28.10023 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 1245.28.10013 Boehringer Ingelheim Investigational Site, Kenosha, Wisconsin
- Argentina (4):
  - 1245.28.54010 Boehringer Ingelheim Investigational Site, Buenos Aires
  - 1245.28.54001 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1245.28.54002 Boehringer Ingelheim Investigational Site, Córdoba
  - 1245.28.54003 Boehringer Ingelheim Investigational Site, Córdoba
- Austria (6):
  - 1245.28.43006 Boehringer Ingelheim Investigational Site, Graz
  - 1245.28.43005 Boehringer Ingelheim Investigational Site, Salzburg
  - 1245.28.43001 Boehringer Ingelheim Investigational Site, Vienna
  - 1245.28.43002 Boehringer Ingelheim Investigational Site, Vienna
  - 1245.28.43003 Boehringer Ingelheim Investigational Site, Vienna
  - 1245.28.43004 Boehringer Ingelheim Investigational Site, Vienna
- Canada (20):
  - 1245.28.20074 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1245.28.20077 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1245.28.20075 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1245.28.20084 Boehringer Ingelheim Investigational Site, Langley, British Columbia
  - 1245.28.20082 Boehringer Ingelheim Investigational Site, Grand Falls-Windsor, Newfoundland and Labrador
  - 1245.28.20016 Boehringer Ingelheim Investigational Site, Mount Pearl, Newfoundland and Labrador
  - 1245.28.20079 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 1245.28.20071 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 1245.28.20080 Boehringer Ingelheim Investigational Site, Collingwood, Ontario
  - 1245.28.20083 Boehringer Ingelheim Investigational Site, Greater Sudbury, Ontario
  - 1245.28.20078 Boehringer Ingelheim Investigational Site, Stayner, Ontario
  - 1245.28.20005 Boehringer Ingelheim Investigational Site, Strathroy, Ontario
  - 1245.28.20072 Boehringer Ingelheim Investigational Site, Chicoutimi, Quebec
  - 1245.28.20081 Boehringer Ingelheim Investigational Site, Chicoutimi, Quebec
  - 1245.28.20085 Boehringer Ingelheim Investigational Site, Gatineau, Quebec
  - 1245.28.20043 Boehringer Ingelheim Investigational Site, Longueuil, Quebec
  - 1245.28.20070 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1245.28.20076 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 1245.28.20073 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
  - 1245.28.20021 Boehringer Ingelheim Investigational Site, Trois-Rivières, Quebec
- Colombia (4):
  - 1245.28.57007 Boehringer Ingelheim Investigational Site, Barranquilla
  - 1245.28.57003 Boehringer Ingelheim Investigational Site, Bogotá
  - 1245.28.57005 Boehringer Ingelheim Investigational Site, Bogotá
  - 1245.28.57006 Boehringer Ingelheim Investigational Site, Floridablanca
- Czechia (8):
  - 1245.28.42003 Boehringer Ingelheim Investigational Site, Brno
  - 1245.28.42005 Boehringer Ingelheim Investigational Site, Holice
  - 1245.28.42002 Boehringer Ingelheim Investigational Site, Mladá Boleslav
  - 1245.28.42008 Boehringer Ingelheim Investigational Site, Prague
  - 1245.28.42001 Boehringer Ingelheim Investigational Site, Slaný
  - 1245.28.42007 Boehringer Ingelheim Investigational Site, Slaný
  - 1245.28.42004 Boehringer Ingelheim Investigational Site, Uherské Hradiště
  - 1245.28.42006 Boehringer Ingelheim Investigational Site, Zlín
- Finland (4):
  - 1245.28.72001 Boehringer Ingelheim Investigational Site, Helsinki
  - 1245.28.72004 Boehringer Ingelheim Investigational Site, Joensuu
  - 1245.28.72003 Boehringer Ingelheim Investigational Site, Oulu
  - 1245.28.72002 Boehringer Ingelheim Investigational Site, Pori
- Hong Kong (3):
  - 1245.28.85201 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1245.28.85207 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1245.28.85202 Boehringer Ingelheim Investigational Site, Kowloon
- India (13):
  - 1245.28.91206 Boehringer Ingelheim Investigational Site, Ahmedabad
  - 1245.28.91202 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.28.91204 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.28.91205 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.28.91208 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.28.91201 Boehringer Ingelheim Investigational Site, Chennai
  - 1245.28.91213 Boehringer Ingelheim Investigational Site, Chennai
  - 1245.28.91203 Boehringer Ingelheim Investigational Site, Hyderabad
  - 1245.28.91211 Boehringer Ingelheim Investigational Site, Kolkata
  - 1245.28.91210 Boehringer Ingelheim Investigational Site, Mangalore
  - 1245.28.91212 Boehringer Ingelheim Investigational Site, New Delhi
  - 1245.28.91207 Boehringer Ingelheim Investigational Site, Pune
  - 1245.28.91209 Boehringer Ingelheim Investigational Site, Uttar Pradesh
- Italy (8):
  - 1245.28.39021 Boehringer Ingelheim Investigational Site, Cagliari
  - 1245.28.39022 Boehringer Ingelheim Investigational Site, Chieri (to)
  - 1245.28.39016 Boehringer Ingelheim Investigational Site, Lucca
  - 1245.28.39018 Boehringer Ingelheim Investigational Site, Milan
  - 1245.28.39019 Boehringer Ingelheim Investigational Site, Milan
  - 1245.28.39017 Boehringer Ingelheim Investigational Site, Monserrato (ca)
  - 1245.28.39023 Boehringer Ingelheim Investigational Site, Rimini
  - 1245.28.39020 Boehringer Ingelheim Investigational Site, Salerno
- Malaysia (8):
  - 1245.28.60003 Boehringer Ingelheim Investigational Site, Johor Bahru
  - 1245.28.60006 Boehringer Ingelheim Investigational Site, Kelantan
  - 1245.28.60005 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 1245.28.60009 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 1245.28.60004 Boehringer Ingelheim Investigational Site, Kuala Pahang
  - 1245.28.60007 Boehringer Ingelheim Investigational Site, Perak
  - 1245.28.60010 Boehringer Ingelheim Investigational Site, Pulau Pinang
  - 1245.28.60001 Boehringer Ingelheim Investigational Site, Selangor Darul Ehsan
- Mexico (4):
  - 1245.28.52006 Boehringer Ingelheim Investigational Site, Aguascalientes
  - 1245.28.52008 Boehringer Ingelheim Investigational Site, Cuautla
  - 1245.28.52009 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1245.28.52007 Boehringer Ingelheim Investigational Site, México
- Netherlands (3):
  - 1245.28.31008 Boehringer Ingelheim Investigational Site, 's-Hertogenbosch
  - 1245.28.31020 Boehringer Ingelheim Investigational Site, Losser
  - 1245.28.31014 Boehringer Ingelheim Investigational Site, Rotterdam
- Norway (3):
  - 1245.28.47002 Boehringer Ingelheim Investigational Site, Hønefoss
  - 1245.28.47001 Boehringer Ingelheim Investigational Site, Oslo
  - 1245.28.47003 Boehringer Ingelheim Investigational Site, Sandefjord
- Philippines (9):
  - 1245.28.63016 Boehringer Ingelheim Investigational Site, Cavite City
  - 1245.28.63013 Boehringer Ingelheim Investigational Site, Cebu City
  - 1245.28.63020 Boehringer Ingelheim Investigational Site, Jaro Iloilo City
  - 1245.28.63004 Boehringer Ingelheim Investigational Site, Manila
  - 1245.28.63015 Boehringer Ingelheim Investigational Site, Manila
  - 1245.28.63012 Boehringer Ingelheim Investigational Site, Pasig
  - 1245.28.63011 Boehringer Ingelheim Investigational Site, Quezon City
  - 1245.28.63010 Boehringer Ingelheim Investigational Site, Tacloban City
  - 1245.28.63014 Boehringer Ingelheim Investigational Site, Tagbilaran City, Bohol
- Portugal (4):
  - 1245.28.35006 Boehringer Ingelheim Investigational Site, Amadora
  - 1245.28.35002 Boehringer Ingelheim Investigational Site, Lisbon
  - 1245.28.35012 Boehringer Ingelheim Investigational Site, Porto
  - 1245.28.35016 Boehringer Ingelheim Investigational Site, Vila Nova de Gaia
- South Africa (10):
  - 1245.28.76019 Boehringer Ingelheim Investigational Site, Boksburg North
  - 1245.28.76018 Boehringer Ingelheim Investigational Site, Bryanston
  - 1245.28.76016 Boehringer Ingelheim Investigational Site, Cape Town
  - 1245.28.76017 Boehringer Ingelheim Investigational Site, Cape Town
  - 1245.28.76012 Boehringer Ingelheim Investigational Site, Durban
  - 1245.28.76015 Boehringer Ingelheim Investigational Site, Durban
  - 1245.28.76013 Boehringer Ingelheim Investigational Site, Krugersdorp
  - 1245.28.76024 Boehringer Ingelheim Investigational Site, Lenasia
  - 1245.28.76023 Boehringer Ingelheim Investigational Site, Lenasia South
  - 1245.28.76014 Boehringer Ingelheim Investigational Site, Pretoria
- Spain (11):
  - 1245.28.34004 Boehringer Ingelheim Investigational Site, Barcelona
  - 1245.28.34011 Boehringer Ingelheim Investigational Site, Barcelona
  - 1245.28.34002 Boehringer Ingelheim Investigational Site, Burjasot
  - 1245.28.34003 Boehringer Ingelheim Investigational Site, Centelles
  - 1245.28.34009 Boehringer Ingelheim Investigational Site, Granada
  - 1245.28.34012 Boehringer Ingelheim Investigational Site, Madrid
  - 1245.28.34013 Boehringer Ingelheim Investigational Site, Madrid
  - 1245.28.34005 Boehringer Ingelheim Investigational Site, Mataró
  - 1245.28.34001 Boehringer Ingelheim Investigational Site, Pineda de Mar
  - 1245.28.34010 Boehringer Ingelheim Investigational Site, San Sebastián de los Reyes
  - 1245.28.34006 Boehringer Ingelheim Investigational Site, Tarrega - Lleida
- Sweden (8):
  - 1245.28.46009 Boehringer Ingelheim Investigational Site, Borås
  - 1245.28.46008 Boehringer Ingelheim Investigational Site, Lund
  - 1245.28.46001 Boehringer Ingelheim Investigational Site, Malmo
  - 1245.28.46005 Boehringer Ingelheim Investigational Site, Örebro
  - 1245.28.46002 Boehringer Ingelheim Investigational Site, Stockholm
  - 1245.28.46006 Boehringer Ingelheim Investigational Site, Stockholm
  - 1245.28.46007 Boehringer Ingelheim Investigational Site, Stockholm
  - 1245.28.46004 Boehringer Ingelheim Investigational Site, Uppsala
- Switzerland (2):
  - 1245.28.41015 Boehringer Ingelheim Investigational Site, Ascona
  - 1245.28.41017 Inselspital Bern, Bern
- Taiwan (5):
  - 1245.28.88004 Boehringer Ingelheim Investigational Site, Changhua
  - 1245.28.88003 Boehringer Ingelheim Investigational Site, Taichung
  - 1245.28.88005 Boehringer Ingelheim Investigational Site, Tainan Hsien
  - 1245.28.88001 Boehringer Ingelheim Investigational Site, Taipei
  - 1245.28.88002 Boehringer Ingelheim Investigational Site, Taipei Hsien
- Thailand (4):
  - 1245.28.66006 Boehringer Ingelheim Investigational Site, Bangkok
  - 1245.28.66007 Boehringer Ingelheim Investigational Site, Bangkok
  - 1245.28.66004 Boehringer Ingelheim Investigational Site, Muang District
  - 1245.28.66008 Boehringer Ingelheim Investigational Site, Nakhonratchasima
- United Kingdom (16):
  - 1245.28.44006 Boehringer Ingelheim Investigational Site, Addlestone
  - 1245.28.44020 Boehringer Ingelheim Investigational Site, Ashford
  - 1245.28.44008 Boehringer Ingelheim Investigational Site, Balham
  - 1245.28.44035 Boehringer Ingelheim Investigational Site, Barnstable
  - 1245.28.44016 Boehringer Ingelheim Investigational Site, Blackpool
  - 1245.28.44021 Boehringer Ingelheim Investigational Site, Bradford-on-Avon
  - 1245.28.44019 Boehringer Ingelheim Investigational Site, Burbage
  - 1245.28.44027 Boehringer Ingelheim Investigational Site, Chestfield, Whitstable
  - 1245.28.44011 Boehringer Ingelheim Investigational Site, Chippenham
  - 1245.28.44022 Boehringer Ingelheim Investigational Site, Chippenham
  - 1245.28.44043 Boehringer Ingelheim Investigational Site, Coventry
  - 1245.28.44025 Boehringer Ingelheim Investigational Site, Doncaster
  - 1245.28.44030 Boehringer Ingelheim Investigational Site, Ely
  - 1245.28.44007 Boehringer Ingelheim Investigational Site, Midsomer Norton
  - 1245.28.44023 Boehringer Ingelheim Investigational Site, Nantwich
  - 1245.28.44017 Boehringer Ingelheim Investigational Site, Whitstable

REFERENCES:
- [Derived] Dennis JM, Young KG, Cardoso P, Gudemann LM, McGovern AP, Farmer A, Holman RR, Sattar N, McKinley TJ, Pearson ER, Jones AG, Shields BM, Hattersley AT; MASTERMIND Consortium. A five-drug class model using routinely available clinical features to optimise prescribing in type 2 diabetes: a prediction model development and validation study. Lancet. 2025 Mar 1;405(10480):701-714. doi: 10.1016/S0140-6736(24)02617-5. Epub 2025 Feb 25. PMID 40020703
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Salem A, Men P, Ramos M, Zhang YJ, Ustyugova A, Lamotte M. Cost-effectiveness analysis of empagliflozin compared with glimepiride in patients with Type 2 diabetes in China. J Comp Eff Res. 2021 Apr;10(6):469-480. doi: 10.2217/cer-2020-0284. Epub 2021 Feb 12. PMID 33576249
- [Derived] Ridderstrale M, Andersen KR, Zeller C, Kim G, Woerle HJ, Broedl UC; EMPA-REG H2H-SU trial investigators. Comparison of empagliflozin and glimepiride as add-on to metformin in patients with type 2 diabetes: a 104-week randomised, active-controlled, double-blind, phase 3 trial. Lancet Diabetes Endocrinol. 2014 Sep;2(9):691-700. doi: 10.1016/S2213-8587(14)70120-2. Epub 2014 Jun 16. PMID 24948511
- [Derived] Ridderstrale M, Svaerd R, Zeller C, Kim G, Woerle HJ, Broedl UC; EMPA-REG H2H-SU trial investigators. Rationale, design and baseline characteristics of a 4-year (208-week) phase III trial of empagliflozin, an SGLT2 inhibitor, versus glimepiride as add-on to metformin in patients with type 2 diabetes mellitus with insufficient glycemic control. Cardiovasc Diabetol. 2013 Sep 5;12:129. doi: 10.1186/1475-2840-12-129. PMID 24007456

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An optional 2-year extension was implemented in this trial through a protocol amendment, which brought the total length of treatment to 4 years. However, some sites did not participate in the 2-year extension, and so considered patients to have completed treatment after 2 years.
Groups:
- Empaglifozin 25 mg: Patients received one Empagliflozin 25 mg tablet and one placebo Glimepiride capsule orally once daily.
  Empagliflozin: 25 mg once daily
  Placebo: Placebo matching Glimepiride
- Glimepiride: Patients received one Glimepiride capsule and one placebo Empagliflozin tablet orally once daily.
  Glimepiride: 1-4 mg once daily
  Placebo: Placebo matching Empagliflozin
Period: Overall Study
Arm/Group | Empaglifozin 25 mg | Glimepiride
Started | 769 | 780
Completed After 2 Years Treatment | 95 | 127
Completed After 4 Years Treatment | 515 | 462
Completed | 610 | 589
Not Completed | 159 | 191
Not completed — Adverse Event | 47 | 51
Not completed — Lack of Efficacy | 4 | 7
Not completed — Non compliant with protocol | 9 | 18
Not completed — Lost to Follow-up | 19 | 20
Not completed — Patient refusal to cont., not due to AE | 45 | 40
Not completed — Not treated | 4 | 0
Not completed — Other not defined above | 31 | 55

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS), All patients randomised, treated with at least one dose of study drug, and with a baseline HbA1c value.
Groups:
- Total: Total of all reporting groups
Arm/Group | Empaglifozin 25 mg | Glimepiride | Total
Number analyzed (Participants) | 765 | 780 | 1545
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (10.3) | 55.7 (10.4) | 55.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 333 | 359 | 692
  Male | 432 | 421 | 853

OUTCOME MEASURES:

1. Secondary Outcome: The Change in Body Weight From Baseline After 104 Weeks of Treatment.
Time Frame: baseline and 104 weeks
Population: FAS (LOCF) - Full Analysis Set (FAS) with Last Observation Carried Forward (LOCF); Values after start of antidiabetic rescue therapy were set to missing and last observation carried forward (LOCF) was used for imputation of missing values.
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Empaglifozin 25 mg | Glimepiride
Number analyzed (Participants) | 765 | 780
kilograms | -3.11 (0.13) | 1.33 (0.13)
Statistical Analysis 1: Comparison: Empaglifozin 25 mg vs Glimepiride; Testing Hierarchy for main analysis (104 weeks): 1. Non-inferiority in HbA1c change from baseline at 104 weeks, 2. Superiority in body weight change from baseline at 104 weeks, 3. Superiority in occurrence of confirmed hypoglycaemic adverse events at 104 weeks, 4. Superiority in HbA1c change from baseline at 104 weeks, 5. Superiority in systolic blood pressure change from baseline at 104 weeks, 6. Superiority in diastolic blood pressure change from baseline at 104 weeks; Test type: Superiority or Other; p < 0.0001, ANCOVA — The superiority tests performed at 104 weeks and the superiority tests performed at 52 weeks both used a nominal significance level of 2.5% to maintain the overall significance level of 5%; ANCOVA with treatment, geographical region, renal function at baseline as fixed effects and baseline weight, baseline HbA1c as linear covariates; Mean Difference (Net) = -4.46, 97.5% CI 2-sided [-4.87 to -4.05], Standard Error of Mean 0.18

2. Primary Outcome: The Change From Baseline in Glycosylated Haemoglobin (HbA1c) After 104 Weeks of Treatment.
Time Frame: Baseline and 104 weeks
Population: FAS (LOCF) - Full Analysis Set (FAS) with Last Observation Carried Forward (LOCF); Values after start of antidiabetic rescue therapy were set to missing and last observation carried forward (LOCF) was used for imputation of missing values.
  .
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Empaglifozin 25 mg | Glimepiride
Number analyzed (Participants) | 765 | 780
percentage of HbA1c | -0.66 (0.03) | -0.55 (0.03)
Statistical Analysis 1: Comparison: Empaglifozin 25 mg vs Glimepiride; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority was tested through a two-sided 97.5% confidence interval for the treatment effect of empagliflozin minus the effect of glimepiride in change from baseline in HbA1c. The null-hypothesis of material inferiority of empagliflozin was rejected if the confidence interval is entirely below the non-inferiority margin 0.3%; p < 0.0001, ANCOVA; ANCOVA with treatment, geographical region, renal function at baseline as fixed effects and baseline HbA1c as linear covariate; Mean Difference (Net) = -0.11, 97.5% CI 2-sided [-0.20 to -0.01], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Empaglifozin 25 mg vs Glimepiride; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0153, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.11, 97.5% CI 2-sided [-0.20 to -0.01], Standard Error of Mean 0.04

3. Secondary Outcome: The Occurrence of Confirmed Hypoglycaemic Events During 104 Weeks of Treatment.
Time Frame: baseline and 104 weeks
Population: Treated set, all patients treated with at least one dose of randomised study drug.
Measure: Number; unit: participants
Arm/Group | Empaglifozin 25 mg | Glimepiride
Number analyzed (Participants) | 765 | 780
participants | 19 | 189
Statistical Analysis 1: Comparison: Empaglifozin 25 mg vs Glimepiride; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Cochran-Mantel-Haenszel test adjusting for baseline HbA1c (<8.5 / >=8.5); Risk Ratio (RR) = 0.102, 97.5% CI 2-sided [0.060 to 0.173]

4. Secondary Outcome: The Change in Systolic Blood Pressure (SBP) From Baseline After 104 Weeks of Treatment.
Time Frame: baseline and 104 weeks
Population: FAS (LOCF-H) - Full Analysis Set (FAS) with Last Observation Carried Forward (LOCF); Values after start of antidiabetic rescue therapy or change of antihypertensive therapy were set to missing and last observation carried forward (LOCF) was used for imputation of missing values.
  .
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Empaglifozin 25 mg | Glimepiride
Number analyzed (Participants) | 765 | 780
mmHg | -3.1 (0.5) | 2.5 (0.5)
Statistical Analysis 1: Comparison: Empaglifozin 25 mg vs Glimepiride; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA with treatment, geographical region, renal function at baseline as fixed effects and baseline SBP, baseline HbA1c as linear covariates; Mean Difference (Net) = -5.6, 97.5% CI 2-sided [-7.0 to -4.2], Standard Error of Mean 0.6

5. Secondary Outcome: The Change in Diastolic Blood Pressure (DBP) From Baseline After 104 Weeks of Treatment.
Time Frame: baseline and 104 weeks
Population: FAS (LOCF-H) - Full Analysis Set (FAS) with Last Observation Carried Forward (LOCF); Values after start of antidiabetic rescue therapy or change of antihypertensive therapy were set to missing and last observation carried forward (LOCF) was used for imputation of missing values.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Empaglifozin 25 mg | Glimepiride
Number analyzed (Participants) | 765 | 780
mmHg | -1.8 (0.3) | 0.9 (0.3)
Statistical Analysis 1: Comparison: Empaglifozin 25 mg vs Glimepiride; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA with treatment, geographical region, renal function at baseline as fixed effects and baseline DBP, baseline HbA1c as linear covariates; Mean Difference (Net) = -2.7, 97.5% CI 2-sided [-3.5 to -1.8], Standard Error of Mean 0.4

6. Secondary Outcome: The Change From Baseline in HbA1c After 52 Weeks of Treatment.
Time Frame: baseline and 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Empaglifozin 25 mg | Glimepiride
Number analyzed (Participants) | 765 | 780
percentage of HbA1c | -0.73 (0.03) | -0.66 (0.03)
Statistical Analysis 1: Comparison: Empaglifozin 25 mg vs Glimepiride; Testing Hierarchy for first interim analysis (52 weeks): 1. Non-inferiority in HbA1c change from baseline at 52 weeks, 2. Superiority in body weight change from baseline at 52 weeks, 3. Superiority in occurrence of confirmed hypoglycaemic adverse events at 52 weeks, 4. Superiority in systolic blood pressure change from baseline at 52 weeks, 5. Superiority in diastolic blood pressure change from baseline at 52 weeks; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.07, 97.5% CI 2-sided [-0.16 to 0.02], Standard Error of Mean 0.04

7. Secondary Outcome: The Change in Body Weight From Baseline After 52 Weeks of Treatment.
Time Frame: baseline and 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Empaglifozin 25 mg | Glimepiride
Number analyzed (Participants) | 765 | 780
kilograms | -3.21 (0.12) | 1.59 (0.11)
Statistical Analysis 1: Comparison: Empaglifozin 25 mg vs Glimepiride; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -4.81, 97.5% CI 2-sided [-5.16 to -4.46], Standard Error of Mean 0.16

8. Secondary Outcome: The Occurrence of Confirmed Hypoglycaemic Events During 52 Weeks of Treatment.
Time Frame: baseline and 52 weeks
Population: Treated set, all patients treated with at least one dose of randomised study drug.
Measure: Number; unit: participants
Arm/Group | Empaglifozin 25 mg | Glimepiride
Number analyzed (Participants) | 765 | 780
participants | 12 | 159
Statistical Analysis 1: Comparison: Empaglifozin 25 mg vs Glimepiride; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Cochran-Mantel-Haenszel test adjusting for baseline HbA1c (<8.5 / >=8.5); Risk Ratio (RR) = 0.077, 97.5% CI 2-sided [0.040 to 0.148]

9. Secondary Outcome: The Change in Systolic Blood Pressure (SBP) From Baseline After 52 Weeks of Treatment.
Time Frame: baseline and 52 weeks
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Empaglifozin 25 mg | Glimepiride
Number analyzed (Participants) | 765 | 780
mmHg | -3.6 (0.5) | 2.2 (0.5)
Statistical Analysis 1: Comparison: Empaglifozin 25 mg vs Glimepiride; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 4, analysis 1]; Mean Difference (Net) = -5.8, 97.5% CI 2-sided [-7.3 to -4.4], Standard Error of Mean 0.6

10. Secondary Outcome: The Change in Diastolic Blood Pressure (DBP) From Baseline After 52 Weeks of Treatment.
Time Frame: baseline and 52 weeks
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Empaglifozin 25 mg | Glimepiride
Number analyzed (Participants) | 765 | 780
mmHg | -1.9 (0.3) | 1.0 (0.3)
Statistical Analysis 1: Comparison: Empaglifozin 25 mg vs Glimepiride; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Net) = -2.8, 97.5% CI 2-sided [-3.7 to -2.0], Standard Error of Mean 0.4

ADVERSE EVENTS:
Time Frame: Up to 4 years.
Description: All adverse events (AE), serious and non-serious, occurring during the course of the clinical trial were collected, documented, and reported to the sponsor by the investigator on the appropriate case report form (CRF) or serious adverse event (SAE) reporting forms.
Groups:
- Empa 25mg: Patients received one Empagliflozin 25 mg tablet and one placebo Glimepiride capsule orally once daily. Empagliflozin: 25 mg once daily Placebo: Placebo matching Glimepiride
Arm/Group | Empa 25mg | Glimepiride
Serious Adverse Events (participants affected / at risk) | 161/765 | 153/780
Other Adverse Events (participants affected / at risk) | 580/765 | 637/780
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Empa 25mg (N=765) | Glimepiride (N=780)
Gastroenteritis (Infections and infestations) | 4 | 0
Cellulitis (Infections and infestations) | 3 | 0
Diverticulitis (Infections and infestations) | 3 | 0
Viral infection (Infections and infestations) | 3 | 0
Bronchitis (Infections and infestations) | 0 | 2
Erysipelas (Infections and infestations) | 1 | 2
Post procedural infection (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 1 | 2
Abscess limb (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Cystitis escherichia (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Hepatitis E (Infections and infestations) | 1 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia legionella (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 1
Salmonellosis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Sialoadenitis (Infections and infestations) | 1 | 0
Tuberculosis gastrointestinal (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic ocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nasal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paranasal sinus benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 3
Goitre (Endocrine disorders) | 1 | 1
Pituitary-dependent Cushing's syndrome (Endocrine disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Adjustment disorder (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Delusional disorder, unspecified type (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 8 | 2
Carpal tunnel syndrome (Nervous system disorders) | 1 | 2
Cerebral haemorrhage (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 2 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 2
Brain stem infarction (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Diabetic coma (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1
Myasthenia gravis (Nervous system disorders) | 1 | 0
Myelopathy (Nervous system disorders) | 1 | 0
Optic neuritis (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Radicular pain (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Thalamic infarction (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 3
Cataract (Eye disorders) | 0 | 2
Diabetic retinopathy (Eye disorders) | 1 | 0
Endocrine ophthalmopathy (Eye disorders) | 0 | 1
Open angle glaucoma (Eye disorders) | 0 | 1
Retinal neovascularisation (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Otosclerosis (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 3 | 8
Acute myocardial infarction (Cardiac disorders) | 1 | 7
Angina unstable (Cardiac disorders) | 4 | 4
Atrial fibrillation (Cardiac disorders) | 4 | 2
Myocardial infarction (Cardiac disorders) | 0 | 3
Myocardial ischaemia (Cardiac disorders) | 1 | 3
Angina pectoris (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Palpitations (Cardiac disorders) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ventricle rupture (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypertensive emergency (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 4 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2
Umbilical hernia (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 1
Anorectal varices (Gastrointestinal disorders) | 0 | 1
Anorectal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Proctitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 4 | 5
Cholecystitis acute (Hepatobiliary disorders) | 1 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 2
Renal failure (Renal and urinary disorders) | 1 | 2
Bladder prolapse (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4 | 3
Menorrhagia (Reproductive system and breast disorders) | 2 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Prostatism (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 2 | 0
Chest pain (General disorders) | 1 | 5
Non-cardiac chest pain (General disorders) | 1 | 2
Cyst (General disorders) | 0 | 1
Hernia (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Sudden death (General disorders) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 8 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 3 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 2
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 2 | 1
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Post procedural constipation (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural headache (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Arrhythmia prophylaxis (Surgical and medical procedures) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Hysterectomy (Surgical and medical procedures) | 1 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 1
Omentectomy (Surgical and medical procedures) | 1 | 0
Oophorectomy bilateral (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empa 25mg (N=765) | Glimepiride (N=780)
Urinary tract infection (Infections and infestations) | 137 | 121
Nasopharyngitis (Infections and infestations) | 90 | 106
Upper respiratory tract infection (Infections and infestations) | 103 | 97
Influenza (Infections and infestations) | 71 | 73
Bronchitis (Infections and infestations) | 34 | 64
Gastroenteritis (Infections and infestations) | 38 | 47
Pharyngitis (Infections and infestations) | 42 | 44
Hypoglycaemia (Metabolism and nutrition disorders) | 41 | 228
Hyperglycaemia (Metabolism and nutrition disorders) | 152 | 227
Dyslipidaemia (Metabolism and nutrition disorders) | 51 | 48
Headache (Nervous system disorders) | 59 | 68
Dizziness (Nervous system disorders) | 62 | 67
Hypertension (Vascular disorders) | 55 | 105
Cough (Respiratory, thoracic and mediastinal disorders) | 53 | 62
Diarrhoea (Gastrointestinal disorders) | 62 | 67
Back pain (Musculoskeletal and connective tissue disorders) | 93 | 90
Arthralgia (Musculoskeletal and connective tissue disorders) | 70 | 86
Pain in extremity (Musculoskeletal and connective tissue disorders) | 51 | 50
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 43 | 43
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 23 | 41

LIMITATIONS AND CAVEATS:
It should be noted that not all patients were followed up for 4 years with regard to the frequencies of adverse events presented up to 4 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.